CLINICAL TRIAL: NCT00198965
Title: Benefits of Sensory-Enhanced Products in Weight Loss and Maintenance
Brief Title: Olestra Containing Foods and Weight Loss and Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Procter and Gamble (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PG1999-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2004-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

INTERVENTIONS:
Behavioral: dietary education
Behavioral: dietary education and provided full fat snack foods
Behavioral: dietary education and provided fat free snack foods

SUMMARY:
This study will be conducted over three phases. Phase I will be a 16-week weight lass phase. Phase II will be a 52-week maintenance phase. Phase III will be a follow-up phase. We will test three diet regimens: 1) an olestra group who will receive a weight-reducing diet that includes olestra-containing products; 2) a triglyceride group who will receive the same weight-reducing diet but with foods made with triglyceride (regular fat); 3) a low-fat group will be instructed to consume a diet made of traditionally low-fat foods that ate available in grocery stores (no olestra foods). These groups will be re-randomized for the maintenance phase and again assigned to one of the three weight loss regimens described above: olestra, triglyceride, or low-fat. In the double-blinded experimental design, groups receiving olestra foods will not be informed of the nutrient contents of the foods or told what fat substitute is used in the preparation. (The consent form will state that a new fat-substitute may be used in the study foods.) During a "run-in" phase, olestra versus regular-fat food sensory and tolerance tests will be conducted.

DETAILED DESCRIPTION:
During Phase I, the three groups will attend mandatory, 1 hour, bi-weekly group meetings. Participants will keep food records for 2 weekdays and 1 weekend day during each 2 week period as well as keeping exercise, snack and sleep logs daily. At each meeting, research staff will collect the completed food records and logs and new forms will be distributed. At weeks 8 and 16 of active weight loss, participants will repeat the assessments (blood tests, body composition, and questionnaires) conducted at baseline to determine treatment-induced changes in each of the dependent measures.

During phase II, all of the groups will participate in group meetings held 1 month after beginning maintenance and quarterly over 52 weeks. Dependent upon group, participants will pick-up foods bi-weekly and body weight will be assessed every 4 weeks. The full battery of assessments will be conducted at 26 weeks and at the end of the maintenance phase at 52 weeks.

Participants will be 180 adults (male and female) between 25 and 50 years of age. The study is designed to answer questions involving an adult population. Participants must be interested in losing weight. Participants must have a body mass index between 30 and 33 because this study is designed to answer questions investigating overweight individuals that are not morbidly obese. Participants with preliminary eligibility, determined via phone screening, will be invited to the clinic for a more in-depth screening including demographic and medical history questionnaires and psychosocial measures. Participants will gibe their consent to provide this information via completing a screening consent form (a separate form from the study consent form). Once this secondary eligibility is determined, a study consent form will be completed, and participants will undergo a baseline screening of physical measures, blood tests (CBC, SMA-20), body composition assessment (via bioelectrical impedance), and complete additional psychosocial questionnaires. Any participants found to be ineligible as a result of these measures will not be permitted to continue in the study, but will be referred for medical care if appropriate. Participants deemed eligible will proceed to the weight loss phase.

ELIGIBILITY:
Inclusion Criteria:

male and female, between 25 and 50 years of age, interested in losing weight, body mass index between 30 and 33, informed consent

Exclusion Criteria:

unwilling to eat study provided foods

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 257
Dates: Start 1999-03; Study Completion 2003-12

PRIMARY OUTCOMES:
weight
blood values
body composition

SECONDARY OUTCOMES:
waist/hip measurements
psychometrics
blood pressure
pulse

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Lutherville, Maryland, United States